CLINICAL TRIAL: NCT04622553
Title: Open-label Extension Study to Evaluate the Long-term Safety and Efficacy of Mexiletine in Paediatric Patients With Myotonic Disorders Who Have Completed the MEX-NM-301 Study.
Brief Title: Open-label Extension Study in Paediatric Patients Who Have Completed the MEX-NM-301 Study.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lupin Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEX-NM-303
Record Dates: First submitted 2020-10-22; First posted 2020-11-10 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Myotonic Disorders
MeSH Terms: conditions — Myotonic Disorders | interventions — Mexiletine

STUDY DESIGN:
Intervention Model Description: The aim of this study is to obtain additional information regarding the long-term safety and efficacy of mexiletine for the symptomatic treatment of myotonia in paediatric subjects who have completed the initial paediatric study MEX-NM-301.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort 1 and 2 (Other): 7 patients aged 12 to < 18 years , inclusive in cohort-1 7 patients aged 6 to < 12 years, inclusive in cohort-2
  Interventions: Drug: Mexiletine

INTERVENTIONS:
Drug: Mexiletine — Patients will be enrolled sequentially into 2 cohorts.
  Cohort 1 - (patients aged 12 to < 18 years):
  approximately 8 weeks - 4 weeks of dose titration period + 4 weeks of maintenance period.
  Cohort 2- (patients aged 6 to < 12 years,):
  approximately 8 weeks - 4 weeks of dose titration period + 4 weeks of maintenance period. Enrolment for Cohort 2 will begin after initial pharmacokinetics (PK), safety and efficacy are confirmed in this population, of patients in Cohort 1
  Other Names: Namuscla ™

SUMMARY:
Open-label Extension Study to Evaluate the Long-term Safety and Efficacy of Mexiletine in Paediatric Patients with Myotonic Disorders Who Have Completed the MEX-NM-301 study.

DETAILED DESCRIPTION:
This is an open-label extension study evaluating the long-term efficacy and safety of mexiletine in paediatric patients with myotonic disorders who have completed the initial parent paediatric study with mexiletine (Protocol No. MEX-NM-301 (PIP Study 4) for children and adolescents aged 6 to < 18 years and who continue to meet the eligibility criteria.

Patients who meet the eligibility criteria and provide consent for this study will be enrolled sequentially by decreasing age groups. Patients aged 12 to < 18 years will enter first as this is the first cohort expected to complete the parent study PIP Study 4 based on top down recruiting. Once initial pharmacokinetics (PK), safety and efficacy are confirmed in this population, patients aged 6 to <12 years will be first enrolled in PIP Study 4 and subsequently this study (PIP Study 7).

Enrolled patients will receive mexiletine at a dose determined in the parent study. Dosing is determined according to body weight and tolerability.

The study includes 9 clinic visits - V1 (baseline), and V2 to V9 every 3 months, approximately, thereafter.

The total duration of study will be 24 months per patient. End-of-treatment (EOT) visit will occur at 24 months or in accordance with the availability of product. The overall study duration would be approximately 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients previously completed the parent study PIP study 4 (MEX-NM-301) and tolerated the Mexiletine in the study.
2. Able and willing to provide assent to study participation and a parent or legal guardian willing to sign written informed consent prior to study entry.
3. Patients continue to meet inclusion criteria of parent study (MEX-NM-301):

   * No significant cardiac abnormalities as determined by a cardiologist's assessment of the ECG and Echocardiogram
   * No history or evidence of any significant liver disorder Laboratory investigations for haematology, biochemistry, and urinalysis at screening are within normal range, or showing no clinically relevant abnormal values, as judged by the Investigator
   * Female patients of childbearing potential must be using an acceptable form of birth control as determined by the Investigator (e.g., oral contraception, implantable, injectable/transdermal hormonal contraception, intrauterine device (IUD), barrier methods), tubal ligation or have a vasectomized partner or are practicing abstinence

Exclusion Criteria:

1. Clinically significant laboratory abnormality, ECG or other clinical findings on physical examination indicative of a clinically significant exclusionary disease as determined by the investigator
2. Any contra-indication to mexiletine (as described in the Namuscla Summary of Product Characteristics [SmPC])

   * Hypersensitivity to the active substance, or to any of the excipients
   * Hypersensitivity to any local anaesthetic
   * Ventricular tachyarrhythmia
   * Complete heart block (i.e., third-degree atrioventricular block) or any heart block susceptible to evolve to complete heart block (first-degree atrioventricular block with markedly prolonged PR interval (≥ 200 ms) and/or wide QRS complex (≥ 120 ms), second-degree atrioventricular block, bundle branch block, bifascicular and trifascicular block),
   * QT interval > 450ms
   * Myocardial infarction (acute or past), or abnormal Q-waves
   * Symptomatic coronary artery disease
   * Heart failure with ejection fraction <50%
   * Atrial tachyarrhythmia, fibrillation or flutter
   * Sinus node dysfunction (including sinus rate < 50 bpm)
   * Co-administration with medicinal products inducing torsades de pointes (class Ia, Ic, III antiarrhythmics): Co-administration of mexiletine and antiarrhythmics inducing torsades de pointes (class Ia: quinidine, procainamide, disopyramide, ajmaline; class Ic: encainide, flecainide, propafenone, moricizine; class III: amiodarone, sotalol, ibutilide, dofetilide, dronedarone, vernakalant) increases the risk of potentially lethal torsades de pointes.
   * Co-administration with medicinal products with narrow therapeutic index
3. Co- administration with antiarrhythmics
4. Any other neurological or psychiatric condition that might affect the assessment of the study measurements
5. Any concurrent illness, or medications which could affect the muscle function
6. Seizure disorder, diabetes mellitus requiring treatment by insulin
7. Pregnant or breastfeeding
8. Concurrent participation in any other clinical trial.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Estimated)
Dates: Start 2021-11-05 (Actual); Primary Completion 2026-01-26 (Estimated); Study Completion 2026-03-12 (Estimated)

PRIMARY OUTCOMES:
Assess the long-term safety and tolerability of mexiletine by AEs | Approximately 24 months
  Assess the long-term safety and tolerability of mexiletine in paediatric patients by number and frequency of AEs/SAEs, throughout the study while on treatment
Assess the long-term safety and tolerability of mexiletine by hand relaxation | Approximately 24 months
  Mean time (in seconds) to relaxation of hand muscles and reduction in relaxation time from the first to the fifth contraction
Assess the long-term safety and tolerability of mexiletine measurement of AESI | Approximately 24 months
  Assess the long-term safety and tolerability of mexiletine in paediatric patients by Incidence of adverse events of special interest (AESI),
Assess the long-term safety and tolerability of mexiletine by changes in ECG | Approximately 24 months
  Assess the long-term safety and tolerability of mexiletine in paediatric patients by changes in ECG assessments from baseline, repeated at each study visit
Assess the long-term safety and tolerability of mexiletine by muscle stiffness | Approximately 24 months
  Score for muscle stiffness (myotonia severity) as self-reported by the patients on a Visual Analog Scale (VAS) or Faces scale

SECONDARY OUTCOMES:
Mean change in VAS | Approximately 24 months
  Mean change in VAS (8 to < 18 years) or Faces (6 to < 8 years) score for severity of muscle stiffness (if not a primary endpoint) pain, weakness and fatigue (every 3 months).
Clinical myotonia assessment | Approximately 24 months
  Mean change in time to open the eyes after forced eye closure as measured on a stopwatch (when eyelid myotonia present)
Mean change in health-related quality-of-life | Approximately 24 months
  Mean change in health-related quality-of-life as measured by the Paediatric Quality of Life (PedsQL) score (secondary endpoint for patients aged 6 years to <18 years; every 6 months).
Clinical Global Impression (CGI) scores | Approximately 24 months
  Clinical Global Impression (CGI) scores (efficacy and tolerability) evaluated by the patient, a parent or proxy and by the investigator. Measured every 6 months
Mean change in Myotonia Behaviour Scale (MBS) scores | Approximately 24 months
  Mean change in Myotonia Behaviour Scale (MBS) scores (for patients aged 6 years to < 18 years; measured every 6 months).
Mean change in time to perform Timed-up and go (TUG) test | Approximately 24 months
  Mean change in time to perform Timed-up and go (TUG) test (patients aged 6 to <18 years only)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Barnérias, MD, Principal Investigator — Hopital universitaire Necker-Enfants Malades
Locations (1):
- Hôpital Necker-Enfants-Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No